CLINICAL TRIAL: NCT03994471
Title: A Study to EvaLuate the EffIcacy and Safety of XyloCore, a Glucose SparIng ExpeRimental Solution, for Peritoneal Dialysis
Brief Title: Efficacy and Safety of XyloCore Peritoneal Dialysis Solution.
Acronym: ELIXIR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Iperboreal Pharma Srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IP-001-18; 2019-004183-21 (EudraCT Number)
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2024-05

CONDITIONS: End Stage Renal Disease
Keywords: peritoneal dialysis; ESRD
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Physioneal 40

STUDY DESIGN:
Intervention Model Description: Randomization will be performed centrally via a web-based system, with stratification according to the presence or absence of diabetes.
Who Masked: Outcomes Assessor
Masking Description: The study cannot be blinded. The assessment of the primary end-point will be performed by a blinded, third party, independent assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XyloCore peritoneal dialysis solution (Experimental): Patients will receive 1, 2 or 3 daily (short-dwell) exchanges with XyloCore of an osmotic strength comparable to their pre-randomization prescription of glucose peritoneal dialysis solution (XyloCore Low, Medium and High Strenght have an osmotic strength comparable to Physioneal, Fixioneal or Dianeal 1.36%, 2.27%, 3.86% glucose, respectively, and Balance, Bicavera, Bicanova or Equibalance with 1.5%, 2.5%, 4.25% glucose, respectively). All patients will receive Extraneal (7.5% Icodextrin) for nocturnal (long-dwell) exchange.
  Interventions: Drug: XyloCore Low Strenght, XyloCore Medium Strenght, XyloCore High Strenght
- Glucose peritoneal dialysis solution (Active Comparator): Patients randomized to glucose solution will continue the 1, 2 or 3 daily (short-dwell) exchanges of Physioneal 40 or 35, Fixioneal 40 or 35 or Dianeal (1.36%, 2.27%, 3.86% glucose), Balance, Bicavera, Bicanova or Equibalance (1.5%, 2.5%, 4.25% glucose) with the same osmotic strength of their pre-randomization prescription. All patients will receive Extraneal (7.5% Icodextrin) for nocturnal (long-dwell) exchange.
  Interventions: Drug: 1.36%, 1.5%, 2.27%, 2.5%, 3.86%, 2.25% Glucose PD Solution

INTERVENTIONS:
Drug: XyloCore Low Strenght, XyloCore Medium Strenght, XyloCore High Strenght — XyloCore Low Strenght: 0.7% Xylitol, 0.5% Glucose, and 0.02% L-carnitine - or - XyloCore Medium Strenght: 1.5% Xylitol, 0.5% Glucose, and 0.02% L-carnitine - or - XyloCore High Strenght: 2.0% Xylitol, 1.5% Glucose, and 0.02% L-carnitine
  Other Names: XyloCore 0.7 or 1.5 or 2.0
  Arms: XyloCore peritoneal dialysis solution
Drug: 1.36%, 1.5%, 2.27%, 2.5%, 3.86%, 2.25% Glucose PD Solution — Physioneal 35 or 40 (including Clear-Flex bag), Fixioneal 35 or 40, Dianeal or Dianeal Low Calcium have 1.36%, 2.27% or 3.86% glucose; Balance, Bicavera, Bicanova or Equibalance have 1.25%, 2.3%, 4.5% glucose.
  Other Names: Physioneal 40 or 35, Fixioneal 40 or 35, Dianeal, Balance, Bicavera, Bicanova, Equibalance
  Arms: Glucose peritoneal dialysis solution

SUMMARY:
Randomized, controlled, parallel groups, open-label, blinded end-point assessment, multicenter study, comparing the effects of a low glucose peritoneal dialysis solution, XyloCore, to glucose solutions (Physioneal, Fixioneal, Dianeal, Balance, Bicavera, Bicanova or Equibalance) only regimen, in patients with End-Stage Renal Disease (ESRD) receiving Continuous Ambulatory Peritoneal Dialysis (CAPD), over a 6-month study period.

DETAILED DESCRIPTION:
Patients should be enrolled if they are receiving 1, 2 or 3 diurnal exchanges of one of the following PD solutions (standard treatment): Physioneal 35 or 40 (including Clear-Flex bag), Fixioneal 35 or 40, Dianeal or Dianeal Low Calcium (1.36%, 2.27% or 3.86% glucose), or Balance, Bicavera, Bicanova or Equibalance (1.5%, 2.3%, 4.25% glucose) - and - one bag of Extraneal (7.5% Icodextrin) for the long-dwell exchange. Patients will be centrally randomized to the investigational product (XyloCore) or the glucose-only PD solution active comparator. Patients randomized to the control group will continue with their prescription of standard treatment with 1, 2 to 3 daily (short-dwell) exchanges of Physioneal, Fixioneal, Dianeal, Balance, Bicavera, Bicanova or Equibalance PD solution. Patients randomized to XyloCore will receive XyloCore Low, Medium or High Strength according to the osmotic strength (glucose concentration) of their prerandomization prescribed PD solution. All patients will keep being prescribed Extraneal (7.5% Icodextrin) for the nocturnal (long-dwell) exchange. The osmotic strength and number of diurnal short dwell exchanges may be modified by the investigator as clinically required. PD prescriptions in both treatment arms should be tailored to reach the minimum target of a total Kt/V of > 1.7 per week throughout the study. A stratified randomization scheme will be employed to ensure balanced allocation across the two treatment groups of patients with diabetes and of patients treated with only 1 diurnal exchange. Randomization will be performed centrally via a web-based system according to a computer-generated randomization list. The study is open-label with blinded evaluator (primary endpoint), without blinding of patients or clinical staff.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Age ≥18 years
2. Diagnosed with ESRD and treated with CAPD in the last 3 months
3. In stable clinical condition during the 3 months before screening as demonstrated by the absence of non-elective hospitalization and major cardiovascular events
4. Have not experienced peritonitis episodes in the last 3 months
5. In treatment with prescribed Extraneal (nocturnal exchange bag solution) for at least 1 month
6. In treatment with 1, 2 or 3 diurnal exchange bag solution of prescribed Phisioneal (including Clear-Flex bag), Fixioneal, Dianeal or Dianeal Low Calcium (1.36%, 2.27% or 3.86% glucose), or Balance, Bicavera, Bicanova or Equibalance (1.25%, 2.3%, 4.5% glucose)
7. Kt/V urea measurement > 1.7 per week at Baseline Visit
8. Followed/treated by the participating clinical Center/Investigator in the last three months
9. Understanding the nature of the study and providing their informed consent to participation.

EXCLUSION CRITERIA:

1. History of drug or alcohol abuse in the six months prior to entering the protocol
2. In treatment with androgens
3. Clinically significant abnormal liver function test (ɣ-GT > 4 times the upper normal limit)
4. Acute infectious conditions (i.e.: pulmonary infection, acute hepatitis, high or low urinary tract infections, renal parenchymal infection, pericarditis, etc)
5. Expected patient's survival shorter than the trial duration
6. History of L-Carnitine therapy or use in the month prior to entering the protocol
7. Have used any investigational drug in the 3 months prior to entering the protocol
8. Female patients who are pregnant or breast-feeding.
9. Female patients of childbearing age (less than 24 months after the last menstrual cycle) who do not use adequate contraception
10. Patients affected by Primary Hyperoxaluria as per known medical therapy
11. Patients with serum levels of uric acid > 7.2 mg/dl (male and postmenopausal women) or > 6.0 mg/dl (premenopausal women)
12. Patients with a major cardiovascular event in the last 3 months
13. Patients with advanced cardiac failure (NYHA 4)
14. Hypersensitivity to any of the constituents of the study IMPs.
15. Any contraindication to the prescribed Peritoneal Dialysis solutions (for long-dwell and short-dwell exchange) as per each product SmPC.
16. Participants with medical history of oxalate or lactate abnormalities considered clinically significant by the investigator.
17. History or evidence of any other medical, neurological or psychological condition that would expose the subject to an undue risk of a significant AE or interfere with study assessments during the course of the trial as determined by the clinical judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Total weekly Kt/Vurea | 24-week
  To measure solutes and calculate peritoneal and renal Kt/V (summing up to total Kt/V), dialysate outflow and urine covering 24 hours will be collected, the volumes will be determined, and a blood sample will be taken

SECONDARY OUTCOMES:
Changes in HbA1c (glycated haemoglobin) | 6 months
  Change from baseline value
Insulin | 6 months
  Changes from the baseline value
LDL cholesterol | 6 months
  Changes from the baseline value
HDL cholesterol | 6 months
  Change from the baseline value
Serum triglycerides | 6 months
  Change from the baseline value
Total cholesterol | 6 months
  Changes from the baseline
Hemoglobin | 6 months
  Changes from the baseline value
EPO requirements | 6 months
  Change from the baseline
Fatigue measured through a validated instrument | 6 months
  Changes from the baseline
Peritoneal ultrafiltration | 6 months
  Changes from baseline
Diuresis (or 24 hours urinary volume) | 6 months
  Changes from baseline
Residual renal function | 6 months
  Changes from baseline - measured as the arithmetic mean of urinary urea and creatinine clearance
Adverse Events | 6 months
  Information about all adverse events, whether volunteered by the patient, discovered by investigator questioning, or detected through physical examination, laboratory test or other means, will be collected, recorded and followed as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Arduino Arduini, MD, Study Director — Iperboreal Pharma; Werner Kleophas, MD, Study Chair — DaVita Deutschland AG
Locations (41):
- Denmark (3):
  - Aalborg University, Aalborg
  - Aarhus University Hospital, Aarhus
  - Zealand University Hospital, Roskilde
- Dialysis Center DaVita, Düsseldorf, Germany
- Italy (19):
  - Ospedale Madonna del Soccorso, Ascoli Piceno
  - Ospedale Santa Maria Annunziata, Bagno a Ripoli
  - Azienda Universitaria Ospedaliera di Bari, Bari
  - ASST Spedali Civili di Brescia, Brescia
  - Ospedale SS. Annunziata, Chieti
  - IRCCS Policlinico San Martino, Genova
  - Ospedale Civile San Salvatore, L’Aquila
  - ASST Fatebenefratelli-Sacco -Ospedale Luigi Sacco, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Universitaria di Modena, Modena
  - AOU Università degli studi della Campania, Napoli
  - Università della Campania L.Vanvitelli, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Ospedale AUSL "Guglielmo da Saliceto", Piacenza
  - Ospedale S.Eugenio, Roma
  - Ospedale C. e G. Mazzoni, San Benedetto del Tronto
  - Azienda Ospedaliera Terni, Terni
  - Ospedale San Giovanni Bosco, Torino
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona
- Spain (8):
  - University Hospital A Coruña Fundación Profesor Novoa Santos, A Coruña
  - Hospital U. Germans Trias i Pujol, Badalona
  - Fundaciòn Puigvert, Barcelona
  - Hospital Universitario Josep Trueta, Girona
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Central De Asturias, Oviedo
- Sweden (2):
  - Halland County Hospital of Halmstad, Halmstad
  - Karolinska University Hospital, Stockholm
- United Kingdom (8):
  - Heartlands Hospital, Birmingham
  - St Luke's Hospital, Bradford
  - University Hospitals Sussex, Brighton
  - Kent and Canterbury Hospital, Canterbury
  - Hammersmith Hospital, London
  - Churchill Hospital, Oxford
  - Sheffield Kidney Institute, Sheffield
  - University Hospitals of North Midlands, Stoke-on-Trent